CLINICAL TRIAL: NCT03114566
Title: Collection and Generation of Antigen-specific T-lymphocyte Cell Lines From Primary, Third-party, Related, and Unrelated Donors
Status: Terminated | Type: Observational
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-211
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: transplant donor; HLA typed; 17-211
MeSH Terms: interventions — Leukapheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consenting healthy donor: Transplant and healthy HLA typed donors
  Interventions: Other: Leukapheresis

INTERVENTIONS:
Other: Leukapheresis — Blood is removed together with an anticoagulant from a vein and separated into white cell rich and red cell rich fractions by centrifugation. The white cells are then saved to generate immune cells and the red cells are reinfused back through the donor's vein.

SUMMARY:
The purpose of this study is to obtain lymphocyte collections from normal healthy volunteer donors in order to create Good Manufacturing Practice grade banks of virus-specific and tumor-reactive T-cells of defined HLA type and restricting HLA allele readily available for therapeutic use.

ELIGIBILITY:
Inclusion Criteria:

* Donors must satisfy standards including those set forth by FACT (Foundation for the Accreditation of Cellular Therapy) and the criteria specified in FDA 21 Code of Federal Regulations (CFR) 1271. Specifically, screening for risk factors for communicable disease as well as infectious disease screening by serologic and PCR testing as outlined below. Including testing for IV, Hepatitis B, Hepatitis C, HTLV I and II, CMV, EBV, and toxoplasmosis, westnile virus, syphilis, varicella zoster, and Chagas disease.
* Donors must be typed for HLA-A, B, C, DR and DQ at high resolution.
* Donors accrued at MSKCC must have a hemoglobin value > 10g/dl
* Donors must be capable of undergoing, at least, a single standard 2 blood volume leukapheresis or a donation of one unit of whole blood
* Donors must weight >/= 25 kg

Exclusion Criteria:

* HTLV/HIV (+) or Hepatitis B or C positive donors
* Donors who are pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Transplant donors and healthy HLA typed volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Generation of T-cells | 1 year
  Blood and/or white cell donations will be used for the generation of the T-cells to be used for adoptive immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Prockop, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org